CLINICAL TRIAL: NCT07179211
Title: Relation Between Neutrophil to Lymphocyte Ratio and Peripheral Artery Disease in Regular Hemodialysis Patients at Sohag University Hospital
Brief Title: Peripheral Artery Disease in Regular Hemodialysis Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Gamal Salem, Resident physician in the Department of General Internal Medicine, Sohag University
Other Study IDs: Soh-Med-25-7-19MS
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Months
Biospecimen Retention: Samples Without DNA — CBC CRP Lipid profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent studies have reinforced the association between high NLR and PAD in hemodialysis patients. This highlights the need for further studies to confirm its predictive value and determine optimal cut-off thresholds tailored to local patient populations. Accordingly, the present study aims to investigate the relationship between NLR and the presence of PAD in patients undergoing regular hemodialysis. By establishing this association in a well-defined population, we hope to provide evidence that supports the use of NLR as a simple, cost-effective tool for PAD risk stratification and early intervention

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years.
* Undergoing maintenance hemodialysis for at least 3 months (thrice weekly)
* Able to provide informed consent.
* Willing to undergo clinical and laboratory evaluations, including peripheral vascular assesment

Exclusion Criteria:

* Active infection or sepsis at the time of evaluation

  .* Patients who have a sedimentation rate of more than 60 mm/hour

  *. Known autoimmune or hematologic disorders that may influence leukocyte count.
* Current use of immunosuppressive therapy, corticosteroids, or chemotherapy.5. History of malignancy.6. Patients with incomplete medical records or unable to undergo peripheral vascular assessment.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The present study aims to investigate the relationship between NLR and the presence of PAD in patients undergoing regular hemodialysis. By establishing this association in a well-defined population, we hope to provide evidence that supports the use of NLR as a simple, cost-effective tool for PAD risk stratification and early intervention
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2026-01-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to evaluate the predictive value of the neutrophil-to- lymphocyte ratio (NLR) for the presence of peripheral artery disease (PAD) in patients undergoing regular hemodialysis. | 6months
% of patients with affection in neutrophills to lymphocytes ratio in parient on regular hemodialysis. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided